CLINICAL TRIAL: NCT02759198
Title: A Randomized, Double-blind, Placebo- and Active-Controlled, Multicenter, Phase 2 Trial to Evaluate the Efficacy and Safety of YH23537 in Patients With Osteoarthritis of the Knee
Brief Title: A Clinical Trial of YH23537 in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YH23537-202
Record Dates: First submitted 2016-04-21; First posted 2016-05-03 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- YH23537 (Experimental): YH23537 750/1500/3000mg
  Interventions: Drug: YH23537
- Celebrex (Active Comparator): Celecoxib 200mg
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator): YH23537 Placebo
  Interventions: Drug: YH23537 placebo

INTERVENTIONS:
Drug: YH23537 — Drug: YH23537 750mg Drug: YH23537 1500mg Drug: YH23537 3000mg
  Other Names: YH23537 750mg/1500mg/3000mg
  Arms: YH23537
Drug: Celecoxib — Drug: Celecoxib 200mg
  Other Names: Celecoxib 200mg
  Arms: Celebrex
Drug: YH23537 placebo — Drug: YH23537 750mg placebo Drug: YH23537 1500mg placebo Drug: YH23537 3000mg placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of YH23537 versus celebrex in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Men and women ≥ 40 years of age
* Patients with knee osteoarthritis at one or both knee by ACR

Exclusion Criteria:

* Patients with known or suspected secondary knee osteoarthritis
* Other exclusions applied

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2017-09-26 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in VAS score to assess pain at Week 12 | baseline and week 12

SECONDARY OUTCOMES:
Change From Baseline in VAS score to assess pain at Week 4, 8 | baseline, week 4 and week 8
Change From Baseline in Western Ontario and McMaster Universities Index of Osteoarthritis (WOMAC) score at Week 4, 8, 12 | baseline, week 4, week 8 and week 12
Change From Baseline in WOMAC subgroup(pain, stiffness, difficulty performing daily activities) score at Week 4, 8, 12 | baseline, week 4, week 8 and week 12
Percentage From Baseline in WOMAC responder at Week 4, 8, 12 | baseline, week 4, week 8 and week 12
Percentage of positive response(+1) in Patient Global Impression of Change (PGIC) at Week 12 | week 12
Percentage of positive response(excellent, good and fair response) in Physician's Global Assessment of Response to Therapy (PGART) at Week 12 | week 12

OTHER OUTCOMES:
Quality of life measured by SF-12 at Week 12 | week 12
Percentage of patients who had taken rescue medication at week 12 | week 12
Amount of rescue medication tablets taken following the investigational product | week 12
The number of days taken rescue medication following the investigational product | week 12
Change From Baseline in Kellgren-Lawrence(KL) grading scale to assess the severity of knee osteoarthritis on a plain radiograph at Week 12 | week 12
Change From Baseline in International knee documentation committee(IKDC) score at Week 4, 8, 12 | week 4, 8, 12

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Je Cho, M.D, Ph.D, Study Chair — Kyunghee University Medical Center
Locations (1):
- KyungHee University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No